CLINICAL TRIAL: NCT07030023
Title: How to Diagnose Wire Syndrome ? A Classification Based on Retrospective Studies and Clinical Experience
Brief Title: Diagnosis of Wire Syndrome
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Ondonto03
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Orthodontic Wires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wire syndrome patients
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — Non intervention

SUMMARY:
The Wire Syndrome (WS) refers to aberrant, unexpected, unexplained, or excessive dental movements involving teeth held by an intact post-orthodontic retention wire. Its prevalence ranging from 1.1% to 43%. It is a chronic, progressive pathological process, generally asymptomatic, resulting in a new malocclusion that is not due to relapse or a physiological process, and whose aesthetic and/or functional dento-periodontal consequences are harmful. The causes are multifactorial origin. In the early stages of Wire Syndrome, dental and periodontal consequences are minors. These issues are thought to progressively worsen over time.However, to date, no author has proposed an appropriate diagnostic approach. Indeed, several diagnostic criteria have been reported in the literature, but their hierarchical ranking, in terms of importance and specificity, has yet to be determined.

The main objective of this study is therefore to propose a classification of WS according to its severity, based on a shared framework between periodontists and orthodontists. This classification should, facilitate early detection of the syndrome, and reduce diagnostic delays and therapeutic errors. It should also help clarify prognosis and improve interprofessional collaboration in developing personalized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Presence of fixed orthodontic retention (maxillary and/or mandible)
* Comprehensive documentation available
* Systemically healthy
* Presence or not of a Wire Syndrome

Exclusion Criteria:

* Patient with other orthodontic retention.
* Patient unable to understand french

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who have undergone orthodontic treatment and are currently wearing a fixed orthodontic retainer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Presence of Wire Syndrome | At the inclusion
  The presence of Wire Syndrome was clinically evaluated (based on photographs) under 2 answers "Yes" or "No".
severity classification of Wire Syndrome | At the inclusion
  Severity was categorized into three grades such as minor, moderate, and severe based on dental and periodontal parameters.

SECONDARY OUTCOMES:
Major clinical diagnosis criteria (Fleiss Kappa) | At the inclusion
  Fleiss Kappa coefficient : minimum value : <0 = no aggreeement; maximum value : > 0.8 = almost perfect.
Minor clinical diagnostis criteria (Fleiss Kappa) | At the inclusion
  Fleiss Kappa coefficient : minimum value : <0 = no aggreeement; maximum value : > 0.8 = almost perfect.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France